CLINICAL TRIAL: NCT02242851
Title: Pharmaco-epidemiological Study Describing the Hypertensive Population Treated With Telmisartan and Conditions of Use by Medical Practitioners and Patients
Brief Title: Study Describing the Hypertensive Population Treated With Telmisartan and Conditions of Use by Medical Practitioners and Patients
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 502.450
Record Dates: First submitted 2014-09-16; First posted 2014-09-17 (Estimated); Last update posted 2014-09-17 (Estimated); Status verified 2014-09

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Telmisartan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Hypertensive patients
  Interventions: Drug: Telmisartan

INTERVENTIONS:
Drug: Telmisartan

SUMMARY:
Primary objective: to characterize hypertensive patients treated for at least 1 month with Telmisartan (alone or in combination with other drugs) in order to define the beneficiary population (those actually receiving the treatment).

Secondary objectives:

* to describe the patients' blood pressure values (when self-monitored) and satisfaction with the treatment (ease of use, efficacy, safety) on the basis of a patient self-questionnaire, filled out 4 weeks after consultation.
* to compare the characteristics of the beneficiary population to those of the initial target population defined in the SPC (summary of product characteristics) for Telmisartan

ELIGIBILITY:
Inclusion Criteria:

* Hypertensive patients treated with Telmisartan for at least one month, consulting a medical practitioner (for whatever reason)

Exclusion Criteria:

Ages: 21 Years to 94 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hypertensive patients treated with Telmisartan for at least one month recruited by ceneral practitioners and cardiologists
Sampling Method: Non-Probability Sample
Enrollment: 5018 (Actual)
Dates: Start 2004-09; Primary Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
Characteristics of hypertensive patients | Baseline, after 1 month of treatment
  Questionnaire to determine the beneficiary population

SECONDARY OUTCOMES:
Changes in blood pressure | Up to 1 month
  Self-monitored by patient
Evaluation of patients satisfaction with treatment | Up to 1 month
  Based on a patient 6-point self-questionnaire